CLINICAL TRIAL: NCT06234852
Title: The Effect of Gradual Withdrawal Versus Maintenance of Low-dose Glucocorticoid in Clinically Quiescent Systemic Lupus Erythematosus, a Pilot Randomized Placebo Controlled Trial.
Brief Title: Gradual Withdrawal of Low-dose Glucocorticoid in Clinically Quiescent Systemic Lupus Erythematosus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LUCRA001
Record Dates: First submitted 2024-01-14; First posted 2024-01-31 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Systemic Lupus Erythematosus, SLE
Keywords: Systemic Lupus Erythematosus; Glucocorticosteroid; Flare
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucocorticoid maintenance group (Active Comparator): Maintenance of 5-mg of prednisolone daily over 24 weeks
  Interventions: Behavioral: Glucocorticoid maintenance group
- Glucocorticoid withdrawal group (Placebo Comparator): Gradual withdrawal of daily 5-mg prednisolone to daily 0-mg prednisolone over 20-24 weeks
  Interventions: Behavioral: Glucocorticoid withdrawal group

INTERVENTIONS:
Behavioral: Glucocorticoid withdrawal group — Gradual withdrawal of daily 5-mg prednisolone to daily 0-mg prednisolone over 20-24 weeks
  Arms: Glucocorticoid withdrawal group
Behavioral: Glucocorticoid maintenance group — Daily 5-mg prednisolone over 24 weeks
  Arms: Glucocorticoid maintenance group

SUMMARY:
This study aims compare the flare rate of maintenance versus gradual withdrawal of 5 mg/day prednisone in systemic lupus erythematosus (SLE) patients with clinically quiescent disease.

DETAILED DESCRIPTION:
Glucocorticoids (GCs) remains the mainstay of treatment in SLE. Prolong used of glucocorticoid can be leading to various organ damage, even in low dose (< 7.5 mg/day). The rational of tapering GCs in SLE who achieve remission or low disease activity is still debated. Recent trial showed the abrupt discontinuation of GCs in sustained clinical remission of SLE increased rate of flare. This study aims compare the flare rate of maintenance versus gradual withdrawal of 5 mg/day prednisone over 24 weeks in systemic lupus erythematosus (SLE) patients with clinically quiescent disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged; 20 years
* Diagnosis of SLE according to Systemic Lupus International Collaborating Clinic (SLICC) classification SLE criteria, 2012.
* Achieved clinically quiescent SLE defined as cSLEDAI-2K = 0 for at least 6 months.
* Current treatment regimen including prednisolone 5mg/day. Prednisolone, antimalarials and/or immunosuppressive therapy had to be stable for at least 4 weeks before randomization.

Exclusion Criteria:

* Pregnant or pregnancy planning
* Unable to follow the schedules
* Overlap with other autoimmune disease, except secondary SjS and APS
* Co-morbid with any other condition which required prednisolone treatment
* Documented adrenal insufficiency

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Any flare according any of 3 definitions | 24 weeks
  Flare definition: 1. Clinical SLEDAI 2K (excluding serology) ≥ 4, 2. Increase in SLE-DAS ≥ 1.72, 3. Increase in clinical SLEDAI-2K plus treatment escalation (including with NSAIDS, glucocorticoids (topical or oral), antimalarials, or immunosuppressants.

SECONDARY OUTCOMES:
Any increase in clinical SLEDAI-2K | 24 weeks
  Percentage of participants with any increase in clinical SLEDAI-2K
Any changes in immunology | 24 weeks
  Percentage of participants with the decrease of C3 or C4 by 50% and/or the increase of anti-dsDNA by 25% as compared with baseline
Any increase in damage accrual | 24 weeks
  Percentage of participants with any increase in Systemic Lupus International Collaborating Clinic/American College of Rheumatology Damage Index (SDI) Score.
Changes in quality of life | 24 weeks
  Changes in Score of Systemic Lupus Erythematosus Quality Of Life (SLEQoL) Questionnaire (mean difference)

CONTACTS AND LOCATIONS:
Overall Officials: Rattapol Pakchotanon, M.D., Study Director — Phramongkutklao College of Medicine and Hospital
Locations (1):
- Rheumatic Disease Unit, Department of Internal Medicine, Phramongkutklao Hospital and College of Medicine, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol is to be shared with others. Full data would become available by mid 2025.
Supporting Information: Study Protocol
Time Frame: Mid 2025
Access Criteria: IPD Sharing Access Criteria has not been decided.

REFERENCES:
- [Derived] Niyompanichakarn S, Chaiamnuay S, Narongroeknawin P, Asavatanabodee P, Leosuthamas P, Pakchotanon R. The Effect of Gradual Withdrawal Versus Maintenance of Low-Dose Glucocorticoid in Clinically Quiescent Systemic Lupus Erythematosus, a Pilot Double-Blind Randomised Controlled Trial. Musculoskeletal Care. 2025 Jun;23(2):e70083. doi: 10.1002/msc.70083. PMID 40148251